CLINICAL TRIAL: NCT01263132
Title: Neuropathic Pain Treatment Using F0434 vs. Gabapentin in Patients With Chronic Distal Diabetic Polyneuropathy: A Randomized, Controlled, Double-blind Study
Brief Title: Neuropathic Pain Management
Acronym: M-F0434
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck S.A. de C.V., Mexico (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200057-500
Record Dates: First submitted 2010-12-14; First posted 2010-12-20 (Estimated); Results first posted 2011-10-27 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Diabetic Neuropathies; Polyneuropathies
Keywords: Polyneuropathy; Diabetes Mellitus; Diabetic peripheral neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Polyneuropathies; Diabetes Mellitus | interventions — Gabapentin; Thiamine; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- F0434 (Experimental)
  Interventions: Drug: F0434
- Gabapentin (Active Comparator)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: F0434 — F0434 will be administered orally with an initial dosage of 3 capsules per day divided into 3 doses with a time interval of 8 hours between each dose. The subject will continue with this dosage for one week and afterwards, the initial dosage will be increased from 3 capsules per day divided into 3 doses with the same time interval between doses, until visit 3 (week 2).
  Other Names: Gabapentin with thiamine and cobalamin
  Arms: F0434
Drug: Gabapentin — Gabapentin will be administered orally with an initial dosage of 3 capsules per day divided into 3 doses with a time interval of 8 hours between each dose. The subject will continue with this dosage for one week and afterwards, the initial dosage will be increased from 3 capsules per day divided into 3 doses with the same time interval between doses, until visit 3 (week 2)
  Other Names: Gababion; Gavindo
  Arms: Gabapentin

SUMMARY:
This is a prospective, randomized, double blind, comparative, experimental controlled Phase 3 clinical trial to assess the efficacy, safety and superiority of F0343 (gabapentin combined with B vitamins) compared to gabapentin alone for treating neuropathic pain in subjects with chronic distal diabetic polyneuropathy.

DETAILED DESCRIPTION:
Subjects will be assigned to one of the two arms of the study, after having been deemed eligible during the screening visit in random double-blind design. Subjects will be evaluated for a 4 week period.

OBJECTIVES

* To assess the effects of F0434 and gabapentin alone on neuropathic pain and Quality Of Life (QOL) of subjects with diabetic neuropathy through a current and validated neuropathic pain scale along with the QOL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with diabetes mellitus type 2
* Subjects with a history of neuropathic pain in the last 3 Months
* Men and women in reproductive age with a family planning method
* Subjects aged between 18 to 70 years
* Subjects with glycosylated haemoglobin (HbA1c) greater than 7% and less than 15%
* Subjects that obtain a grade equal or greater than 4 in the visual analogue scale during the screening visit

Exclusion Criteria:

* Subjects diagnosed as being pregnant or in state of lactation
* Subjects with serum creatinine greater than 1.2 or creatinine depuration in 24 hour urine, less than 60mL/min
* Subjects who are receiving treatment with anti-depressants, anti-epileptics, and are taking vitamin B1 and B12 for treatment of neuropathic diabetes
* Subjects who are being pharmacologically treated for epilepsy
* Subjects diagnosed with rheumatic and hepatic disease and diagnosed with neuropathy for other causes
* Subjects with psychological and psychiatric alteration that hinders adequate collaboration in the study
* Subjects with any orthopaedic alteration of any extremity
* Subjects with peripheral artery disease
* Subjects taking more than two neuropathic pain medicines
* Subjects with history of alcohol, cocaine, marijuana or benzodiazepine substance abuse
* Subjects with acid-peptic disease
* Subjects with history of neoplasm of any type

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck S.A. de C.V., Mexico
Locations (1):
- REMEDI Resultados Médicos Desarrollo e Investigación, S.C., Pachuca, Hidalgo, Mexico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 104 participants were recruited for the study, out of which 29 participants were screen failures which were not randomized and did not receive study treatment.
Groups:
- Gabapentin: Gabapentin 300 mg capsule was taken orally with an initial dosage of 3 capsules per day divided into 3 doses with a time interval of 8 hours between each dose for one week; and then dose increased up to 3 weeks as per dosage adjustment schedule.
- MF0434 + Gabapentin: MF0434 and Gabapentin 300 mg capsule was taken orally with an initial dosage of 3 capsules per day divided into 3 doses with a time interval of 8 hours between each dose for one week and then dose increased up to 3 weeks as per dosage adjustment schedule.
Period: Overall Study
Arm/Group | Gabapentin | MF0434 + Gabapentin
Started | 38 | 37
Completed | 38 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | MF0434 + Gabapentin | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (9.7) | 51.1 (9.9) | 51.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Mean Neuropathic Pain Score at Visit 3 (Week 1)
Description: Neuropathic pain score included 10 pain descriptors (intensity, stinging, burning, dull pain, coldness, sensitivity, numbness, depth, superficial and unpleasant) quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable). Questionnaire generated a score in each of the relevant dimensions and a total score of 0-100. Higher score indicated a greater intensity of pain.
Time Frame: Visit 3 (Week 1)
Population: Per Protocol (PP) population included all participants who were randomized and took at least 1 dose of study medication. In this clinical study Intention to treat (ITT) and PP populations were the same.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Gabapentin | MF0434 + Gabapentin
Number analyzed (Participants) | 38 | 37
Units on a Scale | 51.00 (17.39) | 50.70 (16.67)

2. Secondary Outcome: Quality of Life Survey Assessed Using Short Form 36 (SF-36) Questionnaire
Description: SF-36 is a standardized health survey consisting of 36 questions to measure functional health status. Summary scores are calculated using the following 8 dimensions: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The score for a component is obtained by SF-36 algorithm and it is represented as an average of the individual question scores, which are scaled 0 (not functioning) to 100 (highest functioning). Higher scores are indicative of a better health status.
Time Frame: Visit 2 (Baseline) to Visit 6 (Week 4)
Population: PP population included all participants who were randomized and took at least 1 dose of study medication. In this clinical study ITT and PP populations were the same. Two participants in the MF0434 + Gabapentin group had missing values and hence are not included.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Gabapentin | MF0434 + Gabapentin
Number analyzed (Participants) | 38 | 35
Units on a Scale
  Baseline (Visit 2): General SF-36 QoL Index | 53.044 (22.409) | 56.507 (19.523)
  Week 1 (Visit 3): General SF-36 QoL Index | 65.779 (20.882) | 65.610 (18.599)
  Week 2 (Visit 4): General SF-36 QoL Index | 69.531 (18.987) | 74.370 (15.595)
  Week 3 (Visit 5): General SF-36 QoL Index | 73.058 (18.102) | 78.075 (15.819)
  Week 4 (Visit 6): General SF-36 QoL Index | 78.869 (17.010) | 82.331 (15.793)

3. Primary Outcome: Mean Neuropathic Pain Score at Visit 4 (Week 2)
Description: as for outcome 1
Time Frame: Visit 4 (Week 2)
Population: PP population included all participants who were randomized and took at least 1 dose of study medication. In this clinical study ITT and PP populations were the same.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Gabapentin | MF0434 + Gabapentin
Number analyzed (Participants) | 38 | 37
Units on a Scale | 41.24 (16.21) | 36.94 (15.05)

4. Primary Outcome: Mean Neuropathic Pain Score at Visit 5 (Week 3)
Description: as for outcome 1
Time Frame: Visit 5 (Week 3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Gabapentin | MF0434 + Gabapentin
Number analyzed (Participants) | 38 | 37
Units on a Scale | 33.74 (19.54) | 24.86 (13.52)

5. Primary Outcome: Mean Neuropathic Pain Score at Visit 6 (Week 4)
Description: as for outcome 1
Time Frame: Visit 6 (Week 4)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Gabapentin | MF0434 + Gabapentin
Number analyzed (Participants) | 38 | 37
Units on a Scale | 22.08 (18.54) | 17.29 (15.53)

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Gabapentin | MF0434 + Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 22/38 | 23/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=38) | MF0434 + Gabapentin (N=37)
Drowsiness (Nervous system disorders) | 13 | 6
Dizziness (Nervous system disorders) | 12 | 20
Headache (Nervous system disorders) | 3 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Lower Limb Edema (General disorders) | 1 | 2
Viral Rhinopharyngitis (Infections and infestations) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Acute Otitis Media (Infections and infestations) | 0 | 1
Edema (General disorders) | 0 | 1
Widespread Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Pyrosis (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No